CLINICAL TRIAL: NCT05267093
Title: Efficacy of Acupuncture for Patients With Hand Osteoarthritis: a Randomized, Sham-controlled Trial
Brief Title: Acupuncture vs Sham Acupuncture for Hand Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, weiming wang, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-131-KY
Record Dates: First submitted 2022-02-13; First posted 2022-03-04 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Hand Osteoarthritis
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (Experimental): Participants in acupuncture group will receive treatment at bilateral Baxie (EX-UE9), bilateral Houxi (SI3), bilateral Waiguan (TE5) and Ashi points. The acupuncture treatment will last 30mins for each session, 3 sessions a week (ideally every other day) for a succession of 4 weeks.
  Interventions: Procedure: Acupuncture
- Sham acupuncture group (Placebo Comparator): Participants in sham acupuncture group will receive treatment at bilateral Baxie (EX-UE9), bilateral Houxi (SI3), bilateral Waiguan (TE5) and Ashi points. The sham acupuncture treatment will last 30mins for each session, 3 sessions a week (ideally every other day) for a succession of 4 weeks.
  Interventions: Procedure: Sham acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Sterile single-use stainless steel needles (size 0.3 mm × 25 mm) will be utilized. After local skin disinfection with 75% alcohol wipes, acupuncturists will insert needles perpendicularly into the Ashi points to a depth of approximately 2-3 mm; horizontally into the Baxie points toward the wrist to a depth of 5-10 mm; and perpendicularly into Houxi (SI3) and Waiguan (TE5) to a depth of approximately 5-10 mm. The depth of needling will vary based on the participant's body sizes. After insertion, all needles except those in the Ashi points will be manually manipulated to achieve De qi sensations. All the needles will be retained for 30 min and then gently removed. Participants will take acupuncture treatment three times per week for a total of 12 sessions in 4 consecutive weeks.
  Arms: Acupuncture group
Procedure: Sham acupuncture — The sham needles with blunt tips (size 0.3 mm × 25 mm) will be used in the control group. Acupuncturists will gently lift and twist the sham needles to simulate the treatment procedure, thus blinding the patients to the intervention. Acupuncturist will firstly sterilize the areas of acupoints, then apply the adhesive pads on the surface of Ashi points, Baxie points, Houxi (SI3) and Waiguan (TE5) and insert the sham needles without penetrating. The duration and frequency of treatment sessions will be the same as in the acupuncture group.
  Arms: Sham acupuncture group

SUMMARY:
The investigators plan to conduct this multicentered, sham-controlled randomized clinical trial to evaluate the efficacy and safety of acupuncture for clinical symptomatic improvement of hand OA.

DETAILED DESCRIPTION:
Symptomatic hand osteoarthritis (HOA) is estimated to affect 15.9% of women and 8.2% of men in the general population. Since no therapy can completely cure HOA at present, alternative effective therapies are needed. Acupuncture has been an effective treatment to alleviate pain and improve joint motion for patients with knee osteoarthritis according to a considerable amount of research. It is not surprised that acupuncture is effective in treating HOA in clinical practice considering the similar pathogenesis HOA shared with knee osteoarthritis. However, the research on the effects of acupuncture in patients with HOA is very limited. The present study aims to evaluate the efficacy and safety of acupuncture for HOA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as hand OA according to the American College of Rheumatology (ACR) clinical classification criteria
* History of hand OA for at least 3 months before enrollment and history of taking nonsteroidal anti-inflammatory drugs (NSAIDs) to treat hand OA
* Aged 18-80 years
* At least 40 mm in visual analog scale (VAS) on the average pain intensity of the dominant hand over the last 48 hours (patients applying NSAIDs at the screening have to have an increase in pain in the dominant hand of ≥ 20 mm after 1-week washout)
* Posterior-anterior radiographs of the dominant hand shows Kellgren-Lawrence grade 1, 2, or 3 changes in symptomatic joints
* Negative results in both rheumatoid factor and anticyclonic citrullinated peptide
* Able to comply with the study protocol and understand the medical information forms
* Voluntarily sign the informed consent

Exclusion Criteria:

* History or current evidence of secondary OA (due to causes other than a solely degenerative joint disease) or symptomatic OA at additional locations besides the hand(s) requiring treatment, or any painful syndrome of the upper limb which may interfere with evaluation of hand pain;
* History of inflammatory arthritis (such as rheumatoid arthritis (RA) or psoriatic arthritis), hemochromatosis, metabolic, or neuropathic arthropathies;
* History of trauma, dislocation or operation to the hand or arm in the previous 3 months;
* Hand pain and stiffness due to tissue scarring or tendinitis;
* Skin damage or serious skin disorders in the hands;
* Intake of antidepressants, anticonvulsants, vascular or narcotics during the 10 days prior to beginning the study;
* Oral, intramuscular, intra-articular or intravenous corticosteroids, or hyaluronic acid injection within 3 months preceding enrollment;
* Serious uncontrolled medical conditions such as cancer, uncontrolled cardiovascular disorder, severe hepatic/renal insufficiency or coagulation disorder;
* Known phobic to acupuncture or received acupuncture treatment within 4 weeks prior to enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of responders according to the Outcome Measures in Rheumatological Clinical Trials (OMERACT) and Osteoarthritis Research Society International (OARSI) responder criteria. | week 5
  Participants that meet at least one of the following criteria are considered as responders: 1) at least a 50% decrease and change from baseline≥20 in VAS score; 2) at least a 50% decrease and change from baseline≥20 in Australian Canadian Osteoarthritis Hand Index (AUSCAN); 3) at least a 20% decrease and change from baseline≥10 in at least two measurements of VAS score, AUSCAN and global assessment.

SECONDARY OUTCOMES:
The proportion of responders according to the Outcome Measures in Rheumatological Clinical Trials (OMERACT) and Osteoarthritis Research Society International (OARSI) responder criteria. | week 8 and week 16
  Participants that meet at least one of the following criteria are considered as responders: 1) at least a 50% decrease and change from baseline≥20 in VAS score; 2) at least a 50% decrease and change from baseline≥20 in Australian Canadian Osteoarthritis Hand Index (AUSCAN); 3) at least a 20% decrease and change from baseline≥10 in at least two measurements of VAS score, AUSCAN and global assessment.
Change in average overall finger joints pain intensity in the dominant hand over the past 48h from baseline. | week 5, week 8 and week 16
  Pain intensity will be measured using a 0-100 VAS, with 0 indicating no pain and 100 indicating maximal pain.
Change in maximal overall finger joints pain intensity in the dominant hand over the past 48h from baseline. | week 5, week 8 and week 16
  Pain intensity will be measured using a 0-100 VAS, with 0 indicating no pain and 100 indicating maximal pain.
The proportion of participants achieving at least a 15-point reduction in average overall finger joints pain intensity in the dominant hand from baseline | week 5, week 8 and week 16
  Pain intensity will be measured using a 0-100 VAS, with 0 indicating no pain and 100 indicating maximal pain.
Change in Australian Canadian Osteoarthritis Hand Index (AUSCAN) total score, and pain, stiffness and physical function subscales from baseline. | week 5, week 8 and week 16
  The AUSCAN index contains a 15-item scale referring to hand pain (5 items), stiffness (1 item), and function (9 items) during the preceding 48 hours, which is valid, reliable and responsive in patients with hand OA. All items are scaled on a 0-100 VAS (0=none to 100= very severe), with higher scores indicating more severe symptoms/function.
Change in Functional Index for HOA (FIHOA) from baseline. | week 5, week 8 and week 16
  The FIHOA is a patient-reported hand function questionnaire, comprising 10 items with a four-point Likert scale, in which 0 represents "possible without difficulty", 1 indicates "possible with slight difficulty", 2 represents "possible with important difficulty" and 3 indicates "impossible".
Change in the number of self-reported painful joints and painful joints at digital pressure from baseline. | week 5, week 8 and week 16
  All finger joints will be reported spontaneously for the presence of pain by the participants, and examined by a trained research nurse for the presence of pain at digital pressure.
Change in the number of swollen joints from baseline. | week 5, week 8 and week 16
  All soft swollen finger joints count (0-30) will be assessed by a trained research nurse at each study visit.
Change in hand grip strength of the fingers from baseline. | week 5, week 8 and week 16
  Hand grip strength of the fingers of the dominant hand will be tested using a hand dynamometer.
Change in pinch strength of the fingers from baseline. | week 5, week 8 and week 16
  Hand pinch strength of the fingers of the dominant hand will be tested using a Jamar digital pinch gauge respectively.
Change in patient global assessment of improvement from baseline. | immediately after the intervention, week 8 and week 16
  The patients will be asked to respond to the question 'Considering all the ways your hand OA affects you, how have you been during the last 48 h?' on a self-administered 0-100 VAS (0, worst possible, to 100, best possible, in 10-point increments).
Change in quality of life assessed by the World Health Organization Quality of Life abbreviated version (WHOQOL-BREF) from baseline. | week 5, week 8 and week 16
  The WHOQOL-BREF is a 26-item self-report questionnaire rated on a 5-point Likert-type scale with four domains of QOL: physical (seven items), psychological (six items), social (three items), and environment (eight items), plus 2 items representing the general QOL. The four domain scores are scaled in a positive direction with higher scores indicating a higher quality of life.

OTHER OUTCOMES:
Participants' expectations for acupuncture at baseline. | baseline
  At baseline, participants in both groups will be asked to answer the following question: "What do you expect from EA treatment to improve your hand OA?"
Blinding assessment | immediately after the intervention
  All participants will be told before allocation that insertion is deeper in group A (traditional acupuncture) and shallower in group B (modern acupuncture). After treatments finished, they will be asked "Do you think you were in group A (traditional acupuncture) in the past weeks?", the answers are "Yes", "No" or "Unclear".
Self-reported consumption of acetaminophen for hand OA. | during weeks 1-4, weeks 5-8 and weeks 9-16
  The proportion of participants using acetaminophen, and the frequency and total dosage of acetaminophen used will be calculated and assessed.
Safety assessment | during weeks 1-4, weeks 5-8 and weeks 9-16
  Any acupuncture-associated adverse event (AE) such as dizziness, palpitations, local hematomas, or infection, and any other AE irrelevant to acupuncture, will be carefully documented.

CONTACTS AND LOCATIONS:
Overall Officials: Weiming Wang, Ph.D, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Department of Acupuncture and Moxibustion, China Academy of Chinese Medical Sciences Guang'anmen Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data are available on reasonable request. You can send e-mail to us if you have any question
Supporting Information: Study Protocol, SAP
Time Frame: It depends
Access Criteria: It depends

REFERENCES:
- [Derived] Wang W, Shi H, Liu Y, Sun Y, Chen Y, Liu Z. Efficacy and safety of acupuncture for hand osteoarthritis: study protocol for a multi-center, randomized, sham-controlled clinical trial. J Orthop Surg Res. 2023 Feb 6;18(1):89. doi: 10.1186/s13018-023-03570-6. PMID 36747297